CLINICAL TRIAL: NCT00905320
Title: Sutures or No Sutures (SONS)
Brief Title: Hernia Repair With or Without Sutures
Acronym: SONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Don Selzer, Associate Professor of Surgery, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0803-15
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hernia
Keywords: Hernia repair
MeSH Terms: conditions — Hernia | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metallic Fasteners and Sutures (Active Comparator): Laparoscopic ventral hernia repair with mesh fixation using both metallic fasteners and transabdominal sutures
  Interventions: Procedure: Metallic Fasteners and Sutures
- Metallic Fasteners Alone (Experimental): Laparoscopic ventral hernia repair with mesh fixation using metallic fasteners alone
  Interventions: Procedure: Metallic Fasteners Alone

INTERVENTIONS:
Procedure: Metallic Fasteners and Sutures — Subjects will undergo hernia repair with mesh fixation. Fixation involves using metallic fasteners and sutures.
  Other Names: Metallic fasteners and sutures.
  Arms: Metallic Fasteners and Sutures
Procedure: Metallic Fasteners Alone — Subjects will undergo hernia repair with mesh fixation. Fixation involves using metallic fasteners alone.
  Other Names: Metallic fasteners alone for mesh fixation
  Arms: Metallic Fasteners Alone

SUMMARY:
This is a randomized study between two accepted techniques of mesh fixation for laparoscopic hernia repair.

DETAILED DESCRIPTION:
This is a randomized study in which subjects will undergo one or two currently accepted techniques of mesh fixation during laparoscopic ventral hernia repair. Subject will undergo mesh fixation with either trans-abdominal sutures and metallic tacks or metallic tacks only.

Pain will be assessed through week 12, and hernia recurrence will be assessed for 2 years after surgery. Subjects will complete pain questionnaires at baseline, each day during hospital stay, and at follow-up visits at 2, 6, and 12 weeks after discharge. Quality of life questionnaires will be completed at baseline, at discharge from hospital, and during follow-up visits at 2, 6, and 12 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

Demographics:

* Age ≥ 18 years old
* If female, negative pregnancy test

Pre-Operative Findings:

* Presence of an abdominal hernia associated with previous surgical incision
* Midline ventral\incisional hernia demonstrated either on physical examination by investigators or radiologic imaging tests.
* CT scan, MRI, Ultrasound
* No evidence of incarceration, strangulation
* Size of hernia ≥ 4 centimeters or ≤ 20 centimeters (cross-sectional diameter)
* Multiple hernias cumulative size ≤ 20 centimeters in cross-sectional diameter

Exclusion Criteria:

Pre-Operative History:

* Severe medical co-morbidities that prevent safe performance of laparoscopic surgery including coronary artery disease, obstructive pulmonary disease, etc.
* History of the following:

  * Connective tissue or wound healing disorder (e.g. Ehlers-Danlos syndrome)
  * Chronic use (defined as greater than 3 months) of narcotic analgesic for pain other than from the hernia that is intended to be repaired
* Allergy to products used in hernia repair including surgical mesh
* Any abdominal ventral incisional hernia previously repaired with permanent synthetic mesh placed inside the peritoneal cavity
* Loss of abdominal domain (i.e. majority of abdominal organs lie outside confines of the abdominal musculature and fascia)
* Presence of simultaneous intra-abdominal infection
* Simultaneous presence of a bowel obstruction
* History of suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.

Intra-operative Findings:

* Simultaneous performance of another surgical procedure during hernia repair other than acts necessary to complete hernia repair (e.g. cutting of abdominal adhesions)
* Intra-operative identification of full thickness injury to intestine (i.e. enterotomy), liver, bladder, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2016-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Post-op Pain | 12 Weeks
  Short-Form McGill Pain Questionnaire (SFMP)

SECONDARY OUTCOMES:
Hernia recurrence | 2 Years
  CT Scan

CONTACTS AND LOCATIONS:
Overall Officials: Don Selzer, MD, Principal Investigator — Indiana University Department of Surgery
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No